CLINICAL TRIAL: NCT02517632
Title: Impact of a Physical Exercise Program in Cardiopulmonary RehAbilitation In Patients With Chronic Chagas Heart Disease: a Randomized Controlled Trial (PEACH Trial)
Brief Title: Physical Exercise Program in Chronic Chagas Heart Disease
Acronym: PEACH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Evandro Chagas National Institute of Infectious Disease (Other)
Collaborators: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Fernanda de Souza Nogueira Sardinha Mendes, Researcher, Evandro Chagas National Institute of Infectious Disease
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE:38038914.6.0000.5262
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Chagas Disease; Chagas Cardiomyopathy
Keywords: Physical activity; Cardiac rehabilitation
MeSH Terms: conditions — Chagas Disease; Chagas Cardiomyopathy; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The intervention group performed exercise sessions, pharmaceutical and nutritional counceling. The control group had only pharmaceutical and nutritional counceling.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise group (Experimental): This arm will be submitted to a exercise session and counseling from pharmaceutical and nutritional professionals.
  Interventions: Behavioral: Exercise, nutritional and pharmaceutical counceling
- Control group (Other): This arm will have only the counseling from pharmaceutical and nutritional professionals.
  Interventions: Behavioral: Nutritional and pharmaceutical counceling

INTERVENTIONS:
Behavioral: Exercise, nutritional and pharmaceutical counceling — The exercise group will be submitted to a physical exercise intervention protocol performed three times per week, 60 minutes per session, during 6-month period, and a monthly counseling from pharmaceutical and nutritional professionals provided during the follow-up and consisted on general guidance about healthy eating habits for patients with heart failure, mainly sodium and water intake, and medication usage, particularly drug dosage and compliance.
  Arms: Exercise group
Behavioral: Nutritional and pharmaceutical counceling — The control group will be submitted to a monthly counseling from pharmaceutical and nutritional professionals provided during the follow-up and consisted on general guidance about healthy eating habits for patients with heart failure, mainly sodium and water intake, and medication usage, particularly drug dosage and compliance.
  Arms: Control group

SUMMARY:
The aim of this investigation is to evaluate the impact of exercise in a cardiac rehabilitation program on functional capacity, clinical markers, quality of life and biomarkers in patients with chronic chagasic cardiomyopathy.

DETAILED DESCRIPTION:
The present study consisted in a randomized clinical study conducted at the Evandro Chagas National Institute of Infectious Disease (INI), located on Rio de Janeiro, Brazil. INI is a national reference center for treatment and research in infectious diseases and tropical medicine in Brazil, which follows a large cohort of patients with Chagas disease, all of them diagnosed by two simultaneously positive serological tests (enzyme-linked immunosorbent assay and indirect immunofluorescence). Patients included in the study are randomly divided in two groups: intervention and control groups. Safety analysis will be performed by monitoring any symptoms presented during data collection and follow-up study.

One of the potential risks that the patient may experience during the study is a noninvasive test that will be performed on a treadmill in a controlled environment, with the possibility of the appearance of symptoms such as fatigue, dyspnea, chest pain, dizziness, with minimal chances of occurring complications of difficult clinical control. Except for the blood test and the cardiopulmonary exercise test, the other tests to be performed are non-invasive and do not bring any risk to the participant's health. Will be collect 10 ml of blood which will be stored for up to five years for biomarker assessments.

During the exercise sessions, patients will be clinically monitored for decompensation, need for hospitalization and suspend or end the participation on the study. All cases will be individually assessed to determine the reversibility of the clinical status. Those cases will continue to be followed by the assistant staff, offering all the clinical support available in INI.

ELIGIBILITY:
Inclusion Criteria: (1) Chagas disease diagnosis by serology; (2) chronic chagasic cardiomyopathy, with left ventricular ejection fraction <45% or compensated heart failure (3) clinical stability in the last three months, (4) adherence to the ambulatory clinical treatment and (5) age above 18 years.

Exclusion Criteria: (1) pregnancy, (2) neuromuscular limitations, (3) tobacco use, (4) evidence of nonchagasic heart disease, (5) systemic conditions that limits exercise practice or hemodynamic stress tests (6) unavailability to attend three times a week for a minimum of six months, (7) practitioners of regular exercise and (8) claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Functional capacity measured by peak exercise oxygen consumption | Changes from baselint at three and six months
  This measure is taken during a maximal progressive cardiopulmonary exercise test.

SECONDARY OUTCOMES:
Muscle respiratory strength | Changes from baselint at three and six months
  Maximal inspiratory pressure and maximal expiratory pressure (cmH2O)
Body composition (body fat percentage) | Changes from baselint at three and six months
  Measurement of skinfold thickness were taken at the chest, midaxillary, triceps, subscapular, abdomen, suprailiac and thigh sites on the right side of the body while standing in a relaxed position. The sum of these seven skinfold thicknesses was used to estimate body composition by Jackson & Pollock equation.
Cardiac function (maily ejection fraction) | Changes from baselint at three and six months
  Meaured by echocardiography
Laboratorial biomarkers composite | Changes from baselint at three and six months
  Total cholesterol, HDL-cholesterol, LDL-cholesterol, VLDL-cholesterol,triacylglycerol, glucose, glycated hemoglobin, inflammatory cytokines, Brain Natriuretic Peptide and components of oxidative stress.
Quality of life | Changes from baselint at three and six months
  Minnesota Living with Heart Failure questionnaire (MLHFQ). Score ranging from 0 - 105.
24 hours Holter | Changes from baselint at three and six months
  Cardiac rhythm through continuous dynamic ECG
Nutritional assessment | Changes from baselint at three and six months
  By semiquantitative food frequency questionnaire and 24-hour food intake recall.
Pharmaceutical assessment | Changes from baselint at three and six months
  Semi-structured questionnaires, Morisky´s test, Naranjo Algorithm.
Microvascular reactivity | Changes from baselint at three and six months
  Measured by laser speckle flowmetry
Body mass index | Changes from baselint at three and six months
  Measured by the body weight (kg) divided by squared height (in meters).

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Mendes, M.D., Principal Investigator — Evandro Chagas National Institute of Infectious Disease
Locations (1):
- Evandro Chagas National Institute of Infectious Diseases, Oswaldo Cruz Foundation., Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Vieira MC, Mendes FSNS, da Silva PS, da Silva GMS, Mazzoli-Rocha F, de Sousa AS, Saraiva RM, de Holanda MT, Kasal DAB, Costa HS, Borges JP, Reis MS, Rodrigues Junior LF, Hasslocher-Moreno AM, do Brasil PEAA, Mediano MFF. Effect of an exercise-based cardiac rehabilitation program on quality of life of patients with chronic Chagas cardiomyopathy: results from the PEACH randomized clinical trial. Sci Rep. 2024 Apr 8;14(1):8208. doi: 10.1038/s41598-024-58776-3. PMID 38589582
- [Derived] Mendes Fde S, Sousa AS, Souza FC, Pinto VL, Silva PS, Saraiva RM, Xavier SS, Veloso HH, Holanda MT, Costa AR, Carneiro FM, Silva GM, Borges JP, Tibirica E, Pinheiro RO, Lara FA, Hasslocher-Moreno AM, Brasil PE, Mediano MF. Effect of physical exercise training in patients with Chagas heart disease: study protocol for a randomized controlled trial (PEACH study). Trials. 2016 Sep 2;17(1):433. doi: 10.1186/s13063-016-1553-4. PMID 27590681